CLINICAL TRIAL: NCT01602978
Title: Comparison of Pulse Hemoglobin and Pleth Variability Index to Standard Methods of Guiding Intraoperative Fluid and Transfusion Management During Major Surgical Procedures.
Brief Title: Comparison of Pulse Hemoglobin and Pleth Variability Index
Acronym: Pleth
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Collaborators: Masimo Labs (Other)
Responsible Party: Principal Investigator, Davinder Ramsingh, MD, Principal Investigator, Loma Linda University
Other Study IDs: 5100032
Record Dates: First submitted 2012-03-01; First posted 2012-05-21 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Anemia; Fluid Management
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate whether a validated sensor that is able to measure how much oxygen-carrying molecules called hemoglobin using pulse hemoglobin and Pleth Variability Index (PVI)] are in your blood during surgery can help your doctors manage how much fluid and possibly blood you need to get during your surgery. The hope of the study is that the device may provide an early indication you are having bleeding and this may mean you need to be treated with a transfusion. Our current method of checking this is by getting a blood sample for analysis. The investigators hope is that this device may be able to alert the clinician of the need for blood or fluids without a blood draw being needed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be >18 years old;
* must be having a major surgical procedure;
* The pre-operative estimation of blood loss must be at least 15% of the total blood volume

Exclusion Criteria:

* Does subject have hemoglobinopathy;
* cardiac arrhythmias producing irregular rhythms;
* severe pulmonary disease;
* procedures where loss of more that 10 to 15% of total blood volume is unlikely;
* subject refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adults more than 18 years old that are scheduled for a major surgical procedure.
Sampling Method: Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2010-02; Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
The difference between hemoglobin values from the two monitors. | Pulse hemoglobin will be monitored during the surgery from the first arterial blood gas drawn to the last ABG drawn.
  The primary outcome measure is the difference between hemoglobin values from the pulse oximetry device and from the arterial blood gas co-oximeter.

SECONDARY OUTCOMES:
Difference between measures compared to patient characteristics | Start of surgery to end of surgery
  Secondary outcome measures are the size of difference between measures compared to patient characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Davinder Ramsingh, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States